CLINICAL TRIAL: NCT04980287
Title: Right Gastroepiploic Mesentery Metastasis in Advanced Colon Cancer Locating at or Close to the Hepatic Flexure
Brief Title: Mesogastrium Metastasis in Colon Cancer
Status: Recruiting | Type: Observational
Sponsor: Jichao Qin (Other)
Responsible Party: Sponsor-Investigator, Jichao Qin, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20210649
Record Dates: First submitted 2021-07-20; First posted 2021-07-28 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Colon Cancer
Keywords: colon adenocarcinoma; metastasis; right hemi-colectomy
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Complete mesocolic excision is currently recognized as a standard procedure for colon cancer. Controversy remains on the presence of right gastroepiploic mesentery metastasis in patients with colon cancer locating at or close to the hepatic flexure. The investigators design this study in order to define the incidence of mesogastrium metastasis and analyse the safety and surgical outcome in these patients who undergo complete mesocolic excision with right gastroepiploic mesentery resection.

DETAILED DESCRIPTION:
The development of gastrointestinal surgery has passed over three periods: organ resection, radical resection based on vascular blood vessel center and functional radical organ resection based on membrane anatomy. Using high-definition laparoscopy, surgeons could observe the membrane structure that cannot be identified in traditional open surgery. Total mesocolic excision or complete mesocolic excision has been widely recognized in clinical practice.

In 2009, hohenberger et al. proposed the concept of complete mesocolic excision (CME) for the first time. They retrospectively analyzed the data of 1329 patients with colon cancer who underwent radical resection from 1978 to 2002. They found that the 5-year local recurrence rate decreased from 6.5% to 3.6%, and the 5-year survival rate increased from 82.1% to 89.1%.In 2015, Jianping Gong further introduced the anatomy of mesentery, and highlighted that the radical operation of gastrointestinal tumor should not only complete the traditional D2 or D3 lymph node dissection, but also need the complete excision of the mesentery within the right presumed metastatic tumor cells existingbearing range. On the one hand, its clinical significance lies in reducing intraoperative severe complications; On the other hand, better radical operation and due to avoiding "cancer leakage".

Complete mesocolic excision is currently recognized as a standard procedure for colon cancer. According to the theory of membrane anatomy, the right gastroepiploic mesentery and the mesentery of colon are independent which act as separate envelope. As right gastroepiploic mesentery metastases were classified as distant metastaticmetastasis, radical resection of colon cancer under CME combined with resection of the right gastroepiploic mesentery is not appropriate for patients with colon cancer locating at or close to the hepatic flexure. .

Currently, literatures on the surgical methods and boundary of lymph node dissection for colon cancer are all retrospective studies, and lack of RCT evidence. Controversy remains on the presence of mesogastrium metastasis in patients with colon cancer locating at or close to the hepatic flexure. Therefore, the following questions remain to be addressed: will cancer malignant tumors located locating at or close to hepatic flexure or transverse colon close to flexures metastasize to the right gastroepiploic mesentery (including but not limiting No.6 lymph nodes)? The No.6 lymph node metastasis of No.6 lymph nodes in the patients with colon cancer locating at the hepatic flexure have been reported, but whether the " No.6 lymph nodes " were mixed with lymph nodes in the colon mesentery was unknown. The investigators design this study in order to define the incidence of mesogastrium metastasis in colon cancer locating at or close to the hepatic flexure, and analyse analyze the safety and surgical outcome in these patients undergoing complete mesocolic excision plus right gastroepiploic mesentery resection.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* American Society of Anesthesiologists (ASA) score I to III
* A biopsy proven histological diagnosis of colorectal carcinoma
* Preoperative staging cT2-4aN0M0 or cTanyN+M0
* tumor located at hepatic flexure or transverse colon close to flexures
* Undergoing complete mesocolic excision with right gastric mesentery resection
* Patients have to be aware of the aim of the trial, and have signed the informed consent.

Exclusion Criteria:

* Synchronous colorectal carcinoma
* Clinical evidence of metastasis
* History of colorectal cancer or other malignant tumors
* Preoperative staging cT1N0 or cT4bNany
* Emergency procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the department of GI Surgery of Tongji Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
metastasis rate | an average of 1 year
  the incidence of gastric mesentery metastasis

SECONDARY OUTCOMES:
intraoperative complication | an average of 1 year
  intraoperative complication of complete mesocolic excision plus right gastroepiploic mesentery resection
postoperative complication | an average of 1 year
  postoperative complication of complete mesocolic excision plus right gastroepiploic mesentery resection
3-year DFS | an average of 3 years
  3-year disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No